CLINICAL TRIAL: NCT01850940
Title: Efficacy and Safety of Tolvaptan in Cirrhotic Patients With Hyponatremia - A Multi-center Prospective Cohort Study
Brief Title: Efficacy and Safety of Tolvaptan in Cirrhotic Patients With Hyponatremia
Acronym: OASIS
Status: Completed | Type: Observational
Sponsor: Beijing Friendship Hospital (Other)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Jia Ji-Dong, Direcror of the Liver Research Center, Beijing Friendship Hospital
Other Study IDs: OASIS
Record Dates: First submitted 2013-04-01; First posted 2013-05-10 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Liver Cirrhosis; Hyponatremia
Keywords: Cirrhotic Patients; Hyponatremia; tolvaptan
MeSH Terms: conditions — Liver Cirrhosis; Hyponatremia | interventions — Tolvaptan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Tolvaptan Group: Tolvaptan,qd, po
  Interventions: Drug: Tolvaptan
- Conventional therapy: control group:Conventional therapy without tolvaptan
  Interventions: Other: conventional thearpy

INTERVENTIONS:
Drug: Tolvaptan — Tolvaptan (OPC-41061) is a benzazepine derivative synthesized by Otsuka Pharmaceutical Company, Ltd. Tolvaptan was approved for the treatment of specific forms of hyponatremia by the United States (US) Food and Drug Administration (FDA) in May 2009, the European Medicines Agency on Aug 2009, Japan (Oct 2010), China (Sep 2011) and Korea (Sep 2011). Tolvaptan was approved for the adjunct treatment of volume overload in heart failure by the Japanese Ministry of Health, Labour, and Welfare (MHLW) in Oct 2010. It is also being developed for the treatment of autosomal dominant polycystic kidney disease (ADPKD), and for the treatment of hepatic edema.
  Other Names: OPC-41061
  Groups: Tolvaptan Group
Other: conventional thearpy — conventional therapy with salt limitation ,et al
  Other Names: basic therapy
  Groups: Conventional therapy

SUMMARY:
This is a phase IV, open-label, prospective cohort study for 7 days.The recommended starting dose of tolvaptan is 15 mg daily orally. The dose may be titrated on the next day at 15 mg intervals up to 60 mg daily according to the serum sodium level response.Serum sodium level, change in sodium level from baseline, quality of life (EQ-5D-3L), change in body weight, edema, renal function, mortality and liver-related complications on day 7 and day 30 to evaluate the efficacy of tolvaptan in cirrhotic patients with hyponatremia.

DETAILED DESCRIPTION:
Tolvaptan is an effective treatment for hyponatremia. However, cirrhotic patients were underrepresented in previous studies. The pattern of use and efficacy of tolvaptan in real-life clinical practice are currently unknown.The objective of this study is to evaluate the efficacy of tolvaptan in cirrhotic patients with hyponatremia. The secondary objective is to evaluate the short- to intermediate-term safety of tolvaptan in cirrhotic patients.This will be a phase IV, open-label, prospective cohort study for 7 days. Although not mandatory, study subjects are encouraged to undergo follow-up assessments at 1 month.Subjects will be evaluated at designated time points after initiation of therapy. The primary efficacy endpoint is the proportion of subjects with normal serum sodium level (135-145 mmol/l) on day 7. The secondary efficacy endpoints are serum sodium level, change in sodium level from baseline, quality of life (EQ-5D-3L), change in body weight, edema, renal function, mortality and liver-related complications on day 7 and day 30.

ELIGIBILITY:
Inclusion criteria:

1. Age no less than 18 years;
2. Confirmed cirrhosis by histology or radiological features of cirrhosis and clinical features of portal hypertension;
3. Serum sodium level less than 135 mmol/L;
4. Inpatients.

Exclusion criteria:

1. Clinical features of hypovolemia;
2. Systolic blood pressure less than 90 mmHg;
3. Life expectancy less than one month;
4. History of variceal bleeding in the last six months;
5. Hepatic encephalopathy or peritonitis in the last two weeks;
6. Serum creatinine more than 3.5 mg/dl;
7. Severe cardiopulmonary disease;
8. Urinary tract obstruction.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population of this study will be patients with established cirrhosis and hyponatremia.
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2013-01; Primary Completion 2014-09 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
the proportion of subjects with normal serum sodium level (135-145 mmol/l) | day 7
  evaluate the efficacy of tolvaptan in cirrhotic patients with hyponatremia

SECONDARY OUTCOMES:
change in sodium level from baseline | day 7 and day 30
  evaluate the efficacy of tolvaptan in cirrhotic patients with hyponatremia
quality of life (EQ-5D-3L) | day 7 and day 30
  evaluate the efficacy of tolvaptan in cirrhotic patients
change in body weight | day 7 and day 30
  evaluate the efficacy of tolvaptan in cirrhotic patients with hyponatremia
edema | day 7 and day 30
  evaluate the efficacy of tolvaptan in cirrhotic patients with hyponatremia
renal function | day 7 and day 30
  evaluate the short- to intermediate-term safety of tolvaptan in cirrhotic patients
mortality and liver-related complications | day 7 and day 30
  evaluate the short- to intermediate-term safety of tolvaptan in cirrhotic patients

CONTACTS AND LOCATIONS:
Overall Officials: Dong J Jia, doctor, Study Director — Beijing Friendship Hospital
Locations (19):
- China (19):
  - Beijing Ditan Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Youan Hospital, Beijing, Beijing Municipality
  - Shanghai Renji Hospital, Beijing, Beijing Municipality
  - 302 Military Hospital Integrative Medicine, Beijing, Beijing Municipality
  - 302 Military Hospital Liver Failure Center, Beijing, Beijing Municipality
  - The Third Affiliated Hospital of Sun Yat-sen University, Guangdong, Guangdong
  - Guangdong General Hospital, Guangdong, Guangdong
  - Zhujiang Hospital of Southern Medical University, Guangdong, Guangdong
  - Shanghai Shuguang Hospital Affiliated with Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Huashan Hospital, Shanghai, Shanghai Municipality
  - 85 Militay Hospital, Shanghai, Shanghai Municipality
  - Shanghai Xinhua Hospital, Shanghai, Shanghai Municipality
  - Shanghai Putuo District Central Hospital, Shanghai, Shanghai Municipality
  - Shanghai Changhai Hospital, Shanghai, Shanghai Municipality
  - Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality

REFERENCES:
- [Result] Kim WR, Biggins SW, Kremers WK, et al. Hyponatremia and mortality among patients on the liver-transplant waiting list. N Engl J Med 2008;359:1018-26. Wong VW, Chim AM, Wong GL, et al. Performance of the new MELD-Na score in predicting 3-month and 1-year mortality in Chinese patients with chronic hepatitis B. Liver Transpl 2007;13:1228-35. Serste T, Gustot T, Rautou PE, et al. Severe hyponatremia is a better predictor of mortality than MELDNa in patients with cirrhosis and refractory ascites. J Hepatol 2012;57:274-80. Sanyal AJ, Bosch J, Blei A, et al. Portal hypertension and its complications. Gastroenterology 2008;134:1715-28. Schrier RW, Gross P, Gheorghiade M, et al. Tolvaptan, a selective oral vasopressin V2-receptor antagonist, for hyponatremia. N Engl J Med 2006;355:2099-112. Gheorghiade M, Gattis WA, O'Connor CM, et al. Effects of tolvaptan, a vasopressin antagonist, in patients hospitalized with worsening heart failure: a randomized controlled trial. JAMA 2004;291:1963-71. Cardenas A, Gines P, Marotta P, et al. Tolvaptan, an oral vasopressin antagonist, in the treatment of hyponatremia in cirrhosis. J Hepatol 2012;56:571-8.